CLINICAL TRIAL: NCT05440500
Title: Reliability and Validity Study of Urdu Translation of Western Ontario Shoulder Instability Index in Patients With Shoulder Instability
Brief Title: Reliability and Validity of Urdu Translation of Western Ontario Shoulder Instability Index
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0291
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Instability, Joint
Keywords: Western Ontario Shoulder Instability Index; Urdu Version; Reliability; Validity; Shoulder Instability; Walch-Duplay Score
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to translate Western Ontario Shoulder Instability Index into Urdu and test its authenticity and coherence among the Pakistani community with Shoulder instability.

Also check its correlation with Disability of Arm, Shoulder, and Hand Questionnaire, Rowe score , Walch-Duplay score and Visual Analogue Scale.

DETAILED DESCRIPTION:
The original English version of the Western Ontario Shoulder Instability Index will be translated and culturally adapted .Among Shoulder Instability population, Western Ontario Shoulder Instability Index will provided to 90 participants which will be choose through convenience sampling technique . This sampling method based on pre-defined inclusion and exclusion criteria .To check intra-observer reliability of the final Urdu Translation of Western Ontario Shoulder Instability Index, Disability of Arm, Shoulder, and Hand Questionnaire, Walch-Duplay score, Rowe score and Visual Analogue Scale questionnaires will be filled at the same day by two observers for test inter-observers assessment second application will be applied after 35 minutes of first application. Third assessment will be performed after seven days by first observer. Data will be entered and analyzed by using Statistical Package of Social Sciences Version 24 . Internal consistency will be analyzed with Cronbach's alpha value . Intra-class correlation coefficient will be used to check retest reliability. Urdu Translation of Western Ontario Shoulder Instability Index will be evaluated for content validity ,construct validity ,criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female both patients.
* Pursuing one or more incidences of dislocation, with or without surgical stabilization.
* Participants with glenohumeral joint instabilities.
* Patients between the ages of 20 and 60 who are interested in participating.

Exclusion Criteria:

* History or presence of ;
* The presence of a disease other than the shoulder (osseous, tendinous, vascular,
* inflammatory, radicular, muscular, and so on).
* Shoulder surgery except perhaps surgical stabilization.
* The patient's unwillingness to engage in the study, as well as his or her lack of understanding or fill the questionnaires.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population of Pakistanis with shoulder instability will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability Index | 1st day
  Western Ontario Shoulder Instability Index is an instrument which is used to find out outcomes of shoulder instability treatment . These measures has been used in acute and rehabilitation settings The Western Ontario Shoulder Instability Index covers community based functional activities which are useful for the patients of shoulder instability . It consists of twenty one items related to pain and Activities of Daily Livings
Rowe Score | 1st day
  The Rowe score was divided into two categories based on whether or not widespread ligament laxity was present. The Rowe score is divided into three categories: instability, range of motion, and function.
Disabilities Of Arm, Hand & Shoulder Questionnaire | 1st day
  Disabilities Of Arm, Hand & Shoulder Questionnaire is required for a thorough evaluation of diseases affecting various parts of the arm, as well as for research investigations. It consists of thirty Questions related to pain and Activities of Daily Livings.
Walch-Duplay Score | 1st day
  To measure clinical result, the Walch-Duplay score, which was influenced by the Rowe rating scale, takes into consideration both subjective and objective data: stability, pain, sport level recovery, mobility. It is not self-administered. It consists of four questions for assessment.
Visual Analogue Scale | 1st day
  The Visual Analogue Scale was created to represent the concept of a fundamental continuity. A Visual Analogue Scale is typically a straight stripe measuring 100 mm long, with word descriptions for each end. The patient draws a line through the spot on the line which they believe best describes their present state. The Visual Analogue Scale score is calculated by calculating in millimeters as from the line's left side to the point marked by that of the patient. It usually ranges from "0" indicating "no pain" to the "10" indicating "worst pain".

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No